CLINICAL TRIAL: NCT06237322
Title: An Observational Study Comparing RE.DOCTOR Vitals® Software Accuracy
Brief Title: Study of RE.DOCTOR Vitals® Software Accuracy
Acronym: RE-VITAL
Status: Not yet recruiting | Type: Observational
Sponsor: RE.DOCTOR LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: RDCTR51223
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Respiratory Disorder; Cardiovascular Diseases; Diabetes; Pre-Diabetes; Primary Care
MeSH Terms: conditions — Respiration Disorders; Cardiovascular Diseases; Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Healthy: Blood Pressure, Heart Rate and Respiration Rate Measurements:
  Observations will be made using a medically approved blood pressure monitor, Heart Rate Monitor, Respiration Rate Monitor.
  Measurements will be taken at three specific times:
  In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  Measurement:
  Measurements will be taken at three specific times:
  In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  Observations:
  Participants will be guided on the correct use of the glucometer and instructed to note down readings accurately.
- Cardio vascular diseases: Blood Pressure, Heart Rate and Respiration Rate Measurements:
  Observations will be made using a medically approved blood pressure monitor, Heart Rate Monitor, Respiration Rate Monitor.
  Measurements will be taken at three specific times:
  In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  Measurement:
  Measurements will be taken at three specific times:
  In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  Observations:
  Participants will be guided on the correct use of the glucometer and instructed to note down readings accurately.
- Pre-Diabetes: Blood Glucose Measurement:
  Participants will use a medically approved glucometer to measure their blood glucose levels.
  Measurements will be taken at three specific times:
  In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  PPG Data Collection with Mobile App:
  Before each blood glucose measurement, participants will use the RE.DOCTOR Vitals mobile app to collect raw PPG signals.
  Then without closing the app, they use medical device and enter blood glucose data from the glucometer into the app after each measurement.
  Data collection will be initiated by participants clicking the "collect data" button on the mobile app.
  Observations:
  Participants will be guided on the correct use of the glucometer and instructed to note down readings accurately.
- Diabetes I: Blood Glucose Measurement:
  Participants will use a medically approved glucometer to measure their blood glucose levels.
  Measurements will be taken at three specific times:
  In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  PPG Data Collection with Mobile App:
  Before each blood glucose measurement, participants will use the RE.DOCTOR Vitals mobile app to collect raw PPG signals.
  Then without closing the app, they use medical device and enter blood glucose data from the glucometer into the app after each measurement.
  Data collection will be initiated by participants clicking the "collect data" button on the mobile app.
  Observations:
  Participants will be guided on the correct use of the glucometer and instructed to note down readings accurately.
- Diabetes II: Blood Glucose Measurement:
  Participants will use a medically approved glucometer to measure their blood glucose levels.
  Measurements will be taken at three specific times:
  In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  PPG Data Collection with Mobile App:
  Before each blood glucose measurement, participants will use the RE.DOCTOR Vitals mobile app to collect raw PPG signals.
  Then without closing the app, they use medical device and enter blood glucose data from the glucometer into the app after each measurement.
  Data collection will be initiated by participants clicking the "collect data" button on the mobile app.
  Observations:
  Participants will be guided on the correct use of the glucometer and instructed to note down readings accurately.

SUMMARY:
The purpose of this observational trial is to advance digital health monitoring through the analysis of Photoplethysmography (PPG) waveforms collected via RE.DOCTOR Vitals software. The study aims to collect a diverse and extensive dataset of PPG waveforms, alongside traditional physiological measurements, for the purpose of enhancing existing algorithms and machine learning models used in health monitoring. The primary focus is on improving the accuracy and reliability of algorithms in interpreting PPG data to derive meaningful insights into physiological parameters. The main questions it aims to answer are:

* How can extensive datasets of PPG waveforms be utilized to enhance existing algorithms and machine learning models?
* How do correlations between PPG waveforms and key physiological parameters (such as glucose levels, blood pressure, heart rate, respiration rate) contribute to refining algorithms for more accurate and reliable health predictions?

Participants will be asked to:

* Continuously monitor their health using smartphone applications.
* Allow the collection of PPG waveforms in diverse settings.
* Engage in tasks related to monitor health parameters using medically approved devices

DETAILED DESCRIPTION:
1.1 Introduction Physiological parameters, such as glucose levels, blood pressure, blood oxygen, respiration rate, and pulse, are critical indicators of an individual's health. Monitoring these parameters is crucial for early detection and management of various health conditions. Photoplethysmography (PPG) has emerged as a non-invasive and convenient method for capturing real-time cardiovascular information. In the context of this study, the focus is on leveraging PPG data collected through smartphone applications to enhance the performance of existing algorithms and machine learning models.

1.2 Rationale for the Study The rationale for this study lies in the potential of PPG data to contribute significantly to the refinement of algorithms and machine learning models for health monitoring. While existing models have shown promise, collecting more diverse and extensive datasets can address limitations and improve their accuracy and reliability. By understanding the nuances of PPG waveforms in relation to key physiological parameters, the investigators aim to advance the field of digital health and contribute to the development of more effective monitoring solutions.

1.3 Significance of the Study The significance of this observational trial extends to the optimization of health monitoring algorithms. Improving the accuracy of existing models through extensive data collection can lead to more reliable insights into an individual's health status. The study's findings may influence the development of algorithmic solutions for personalized health monitoring, paving the way for more precise and timely interventions based on real-time physiological data.

2. Objectives

2.1 Primary Objective

Primary Objective:

To collect a diverse and extensive dataset of PPG waveforms, alongside traditional physiological measurements, for the purpose of enhancing existing algorithms and machine learning models used in health monitoring. The primary focus is on improving the accuracy and reliability of algorithms in interpreting PPG data to derive meaningful insights into physiological parameters.

Rationale:

The primary objective aligns with the overarching goal of optimizing existing algorithms. By collecting a comprehensive dataset, we aim to provide a robust foundation for refining and training machine learning models, ultimately enhancing their capacity to accurately interpret and correlate PPG waveforms with key physiological parameters.

2.2 Secondary Objectives

Secondary Objectives:

To explore variations in PPG waveforms across diverse demographic groups and health conditions to ensure the generalizability of algorithmic improvements.

To assess the impact of increased data volume on the performance and scalability of existing algorithms.

To validate the optimized algorithms through comparison with traditional physiological measurements and clinical assessments.

To engage participants in the study for feedback on the usability and acceptability of the smartphone application for continuous health monitoring.

Rationale:

The secondary objectives complement the primary goal by addressing specific aspects of algorithmic improvement. Exploring demographic variations ensures that the refined algorithms remain applicable across diverse populations. Assessing the impact of increased data volume and validating against traditional measurements contribute to the overall robustness and reliability of the optimized algorithms.

Following informed consent, participants will be assigned to sub-protocols for the assessment of the RE.DOCTOR Vitals Software. The study aims to evaluate the accuracy and usability of the software in monitoring vital signs and blood glucose.

Recruitment Criteria:

Participants with the capacity to consent may be assigned to one or to more than one cohort.

All individuals will undergo the following measurements:

* Blood Pressure Measurement
* Heart Rate Measurement
* Respiration Rate Measurement
* Blood Oxygen Measurement
* Blood Glucose

Measurement Procedures:

Pre-measurement Observation:

Demographic and medical history questions.

Routine Observations:

Measurements taken using standard clinical equipment. Measurement taken using similar tools (phone app using PPG) PPG signal capture and health parameters estimated (Heart rate, Respiration Rate, Blood Pressure, Blood Oxygen, Blood Glucose) of the participant's finger using the RE.DOCTOR Vitals app during approx 60 seconds.

Blood glucose measurement using standard procedures.

Post-measurement Observation:

Completion of post-measurement observation questions.

Questionnaire:

A subset of participants from both sub-protocols will be asked to complete a questionnaire related to vital sign monitoring, including preferences for RE.DOCTOR Vitals or other technologies.

Overall Study Protocol:

The study comprises two sub-protocols - Sub-protocol A for blood pressure, heart rate, and respiration rate measurements, and Sub-protocol B for blood glucose measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age between 13-80 years.
* Ownership of a smartphone compatible with the designated data collection application.
* Willingness to use the smartphone application for continuous PPG data collection.
* Ability to provide informed consent for participation in the study.
* No known history of conditions or medications that significantly affect PPG waveforms (e.g., severe arrhythmias, use of beta-blockers).
* Healthy individuals and individuals with diagnosed CVD diseases, individuals with diagnosed pre-diabetes, diabetes I, diabetes II

Exclusion Criteria:

* Age outside the specified range of 13-80 years.
* Lack of ownership of a compatible smartphone.
* Inability or unwillingness to use the designated smartphone application for data collection.
* Known history of severe arrhythmias or use of medications affecting cardiovascular function.
* Any condition that, in the judgment of the investigator, may compromise the participant's ability to complete the study.

Ages: 13 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The inclusion criteria are designed to ensure that participants are within a target age range, have access to the required technology, and are willing and able to actively participate in the study. The criteria also aim to exclude individuals with conditions or medications that could potentially confound the relationship between PPG waveforms and physiological parameters.
  Exclusion criteria are defined to ensure the safety and feasibility of participants in the study. Excluding individuals with specific health conditions or medications that could significantly affect PPG waveforms helps maintain the integrity of the data and the validity of the study outcomes.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Systolic and Diastolic Blood Pressure Measurement taken with RE.DOCTOR Vitals Software | Measurements will be taken at three specific times: In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  Systolic and Diastolic Blood Pressure Measurement taken with RE.DOCTOR Vitals Software
Systolic and Diastolic Blood Pressure Measurement taken with medical device | Measurements will be taken at three specific times: In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  Systolic and Diastolic Blood Pressure Measurement taken with medical device
Systolic and Diastolic Blood Pressure Measurement taken with alternate PPG software device | Measurements will be taken at three specific times: In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  Systolic and Diastolic Blood Pressure Measurement taken with alternate PPG software device
Heart Rate Measurement taken with RE.DOCTOR Vitals Software | Measurements will be taken at three specific times: In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  Heart Rate Measurement taken with RE.DOCTOR Vitals Software
Heart Rate Measurement taken with medical device | Measurements will be taken at three specific times: In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  Heart Rate Measurement taken with medical device
Heart Rate Measurement taken with alternate PPG software device | Measurements will be taken at three specific times: In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  Heart Rate Measurement taken with alternate PPG software device
Respiration Rate Measurement taken with RE.DOCTOR Vitals Software | Measurements will be taken at three specific times: In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  Respiration Rate Measurement taken with RE.DOCTOR Vitals Software
Respiration Rate Measurement taken with medical device | Measurements will be taken at three specific times: In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  Respiration Rate Measurement taken with medical device
Respiration Rate Measurement taken with alternate PPG software device | Measurements will be taken at three specific times: In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  Respiration Rate Measurement taken with alternate PPG software device
Blood Oxygen Measurement taken with RE.DOCTOR Vitals Software | Measurements will be taken at three specific times: In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  Blood Oxygen Measurement taken with RE.DOCTOR Vitals Software
Blood Oxygen Measurement taken with medical device | Measurements will be taken at three specific times: In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  Blood Oxygen Measurement taken with medical device
Blood Oxygen Measurement taken with alternate PPG software device | Measurements will be taken at three specific times: In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  Blood Oxygen Measurement taken with alternate PPG software device
Blood Glucose Measurement taken with RE.DOCTOR Vitals Software | Measurements will be taken at three specific times: In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  Blood Glucose Measurement taken with RE.DOCTOR Vitals Software
Blood Glucose Measurement taken with medical device | Measurements will be taken at three specific times: In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  Blood Glucose Measurement taken with medical device
Blood Glucose Measurement taken with alternate PPG software device | Measurements will be taken at three specific times: In the morning after 6-8 hours of sleep. 2 hours after the first meal of the day. Before bedtime.
  Blood Glucose Measurement taken with alternate PPG software device

CONTACTS AND LOCATIONS:
Locations (1):
- Re.Doctor, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: RE.DOCTOR — https://re.doctor